CLINICAL TRIAL: NCT00585442
Title: Effects of Calcitriol (1α, 25-[OH]2 Vitamin D3) on Renin Expression in Hypertensive Patients Without Vitamin D Deficiency
Brief Title: Effects of Vitamin D on Renin Expression in Hypertensive Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of quality data
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, mark munger, Professor, Pharmacotherapy, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22714; 10151812 (Other Grant/Funding Number: American Foundation for Pharmaceutical Education)
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension; Vitamin D Deficiency
MeSH Terms: conditions — Hypertension; Vitamin D Deficiency | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcitriol (Experimental)
  Interventions: Drug: calcitriol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: calcitriol — 1.0 mcg daily
  Other Names: Rocaltrol; 1α, 25-[OH]2 Vitamin D3
  Arms: Calcitriol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The cardiovascular effects of vitamin D therapy (in humans) have been documented only in patients with known vitamin D deficiency or hyperparathyroidism (a surrogate marker of inadequate vitamin D activity). It is unknown whether the cardiovascular benefits of vitamin D therapy extend beyond these patients to the general hypertensive population. We propose to directly measure the effect of vitamin D therapy on plasma renin activity (PRA), plasma renin concentration (PRC), renin transcription (in mononuclear leukocytes), and blood pressure in hypertensive (but otherwise healthy) patients in a randomized, controlled, experimental trial. This will be the first study to assess vitamin D receptor (VDR) biological (PRA, PRC, renin mRNA, and polymorphisms) and hypertensive activity in patients without vitamin D deficiency. We hypothesize that vitamin D inhibition of renin transcription will produce significant reductions in PRA, PRC, renin transcription, inflammatory cytokines, SBP, and DBP, with potential variation by VDR genotype. Such a result may prove to be significant in the treatment of hypertension, as even modest blood pressure reductions (5 mmHg) are associated with a 14% reduction in mortality due to stroke, a 9% reduction in mortality due to CHD, and a 7% overall reduction in all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age > 55 years.
2. Female patients must be postmenopausal, as determined by surgical hysterectomy or 12 month history since last active menstruation
3. Stage I hypertension (JNC VII Criteria): mean systolic blood pressure (mSBP) 140-159 mmHg and mean diastolic blood pressure 90 - 99 mmHg (mDBP)2
4. Provide informed consent

Exclusion Criteria:

1. Serum vitamin D <55 pmol/L
2. Serum calcium >10.5 mg/dL
3. Serum phosphate (inorganic) >5.5 mg/dL
4. Serum parathyroid hormone (PTH) >1.3 pmol/L
5. Vitamin D supplements, calcium supplements, estrogen replacement therapy, corticosteroids (inhaled/oral), or hydroxymethyl glutarate CoA reductase inhibitors (statins) within 30 days prior to randomization
6. Stage II hypertension (JNC VII criteria): mSSBP >160 mmHg or mSDBP >100 mmHg
7. Use of alpha2-agonists, beta-blockers, or more than 2 anti-hypertensive medications at screening
8. Estimated creatinine clearance <30 mL/min by Crockroft-Gault Formula
9. History of heart failure (HF), acute myocardial infarction (AMI), acute coronary syndrome (ACS), transient ischemic attack (TIA), cerebrovascular accident (CVA), peripheral vascular disease (PVD), or known clotting disorder
10. Insulin dependent diabetes mellitus (patients stabilized on oral regimens may be enrolled)
11. History of hypersensitivity reaction to 1α, 25-(OH)2 vitamin D3 (calcitriol)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Compare plasma renin activity (PRA) and plasma renin concentration (PRC) in hypertensive patients (JNC VII stage I) following 14 days treatment with calcitriol (1α, 25-[OH]2 vitamin D3) or matched placebo. | 13 MONTHS (MAY 2007-JUNE 2008)

SECONDARY OUTCOMES:
Compare mononuclear leukocyte renin transcription (mRNA) between calcitriol and matched placebo. | 13 MONTHS (MAY 2007-JUNE 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Munger, PharmD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States